CLINICAL TRIAL: NCT06151002
Title: PD Frontline, Part of RAPSODI GD (Remote Assessment of Parkinsonism Supporting Ongoing Development of Interventions in Gaucher's Disease) to Build an Online Trial-ready Cohort of GBA Genotyped People With Parkinson's
Brief Title: PD Frontline (Part of RAPSODI GD) Remote Assessment of People With Parkinson's
Acronym: PD Frontline
Status: Recruiting | Type: Observational
Sponsor: University College London Hospitals (Other)
Collaborators: Cure Parkinson's (Other)
Responsible Party: Principal Investigator, Anthony Schapira, Professor Anthony Schapira, University College London Hospitals
Other Study IDs: 173275
Record Dates: First submitted 2023-10-11; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Extracted DNA from saliva samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PD Frontline (part of RAPSODI GD) is an online study observational study with the goal of bringing People with Parkinson's to the frontline of research by getting them trial ready. To do this, participants are offered genetic sequencing for the GBA and LRRK2 gene with an at-home saliva collection kit.

DETAILED DESCRIPTION:
PD Frontline is an online one-time questionnaire based study with the purpose of identifying potential candidates for gene targeted trials and observational studies.

Once the questionnaire is completed, the participant is sent a saliva collection kit in the post to provide a sample for genetic testing. The genes tested for are GBA1, the most common risk factor gene for Parkinson's, and LRRK2.

Once tested, the participant is informed of their results and kept up-to-date with any studies or trials for which they may be eligible.

ELIGIBILITY:
Inclusion Criteria:

* Formal diagnosis of Parkinson Disease

Exclusion Criteria:

* Confirmation that the individual carries a GBA variant (GBA positive). These individuals will be referred to sister-study, RAPSODI.
* History of Parkinsonism (progressive supranuclear palsy, multiple system atrophy, traumatic, manganese toxicity, postencephalitic, vascular PD; drug induced PD; corticobasal degeneration)
* Individuals with another neurological disorder including: dementia, movement disorders, and motor neurone disease.
* Individuals on drugs known to be associated with parkinsonism, including neuroleptic agents (Amisulpride, Chlorpromazine Hydrochloride, Flupenthixol, Fluphenazine Hydrochloride, Haloperidol, Methotrimeprazine, Levomepromazine, Olanzapine, Oxypertine, Pericyazine, Perphenazine, Pimozide, Pipotiazine, Prochlorperazine, Promazine Hydrochloride, Reserpine, Risperidone, Sulpiride, Thioridazine, Trifluoperazine, Zuclopenthixol acetate, Zotepine), plus Bupropion, , Lithium, Methyldopa, Metoclopramide and Sodium Valproate).

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Randomly selected population, recruited via established NHS sites and self-referral to the website.
Sampling Method: Non-Probability Sample
Enrollment: 4800 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2025-02-14 (Estimated); Study Completion 2040-08-20 (Estimated)

PRIMARY OUTCOMES:
Genotype of participants | 20 years
  The primary outcome of the study is to genotype the GBA1 gene, obtained with Oxford Nanopore long read sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London (UCL), London, United Kingdom